CLINICAL TRIAL: NCT02559245
Title: Effect of Flixweed and Fig on Irritable Bowel Syndrome With Predominant Constipation: a Single Blind Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Makan Pourmasoumi, MSc Student, Food Security Research Center, Department of Community nutrition, School of Nutrition & Food Sciences, Isfahan University of Medical Sciences, Isfahan, Iran, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: makan.pourmasoumi@gmail.com
Record Dates: First submitted 2015-09-21; First posted 2015-09-24 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Irritable Bowel Syndrome Predominant Constipation

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Ficus carica (Experimental): 45 grams Ficus carica before breakfast and lunch with 1 glass of water every day respectively (total consumption: Ficus carica 90g/d)
  Interventions: Other: Ficus carica
- Descurainia Sophia (Experimental): 30 grams Descurainia Sophia before breakfast and lunch with 1 glass of water every day respectively (total consumption: Descurainia Sophia 60g/d)
  Interventions: Other: Descurainia Sophia
- controled (No Intervention): participants will follow their usual diet

INTERVENTIONS:
Other: Descurainia Sophia
  Arms: Descurainia Sophia
Other: Ficus carica
  Arms: Ficus carica

SUMMARY:
This study evaluates effect of Ficus carica and Descurainia Sophia on irritable bowel syndrome predominant constipation. one-third of patients will receive Ficus carica, another one-third will receive Descurainia Sophia and remained patients only will follow their regular diet for 4 months.

ELIGIBILITY:
Inclusion Criteria:

* patients with irritable bowel syndrome predominant constipation

Exclusion Criteria:

* Subjects with significant cardiovascular, renal, hepatic, pulmonary, endocrine, metabolic, hematologic disorders,
* structural abnormalities of the gastrointestinal tract or
* diseases ⁄conditions that affected bowel transition,
* surgery,
* any prokinetic or laxative drug used during the past month,
* any medication that may affect gastrointestinal motility,
* other therapeutic dietary advice for IBS,
* used Fig or Flixweed during the last month,
* diarrhea,
* pregnancy or
* breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
irritable bowel syndrome constipation predominant symptom | 4 months
  IBS severity score system questionnaires will use for evaluation of IBS-C symptoms at the pre and post-intervention. This tool is validated for use in IBS patients that assess 5 clinically relevant items during past 10-days and including severity of abdominal pain, frequency of abdominal pain, severity of abdominal distention, dissatisfaction with bowel movement and interference of IBS with life in general. Each items was scored with a 100 mm visual analogue scale (VAS).

SECONDARY OUTCOMES:
quality of life in IBS-C patients | 4 months
  quality of life in IBS-C patients were assessed at pre-and post-intervention using a self-report Irritable Bowel Syndrome-Quality of Life Measure (IBS-QoL). It contains 34 items with 8 sub-classification including dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual, and relationships. The sum of response to this items by every subject were average and transform to 0-100 scale. The higher score indicated better quality of life among IBS-C patients.
frequency of defecation and hard stool | 4 months
  frequency of defecation and hard stool was evaluated at baseline and end of every month using the visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: makan pourmasoumi, MSc, Principal Investigator — Food Security Research Center, Isfahan University of Medical Sciences, Isfahan, Iran
Locations (1):
- Gastrointestinal Research Center, Isfahan, Iran